CLINICAL TRIAL: NCT07176962
Title: A Cell-free DNA Methylation Liquid Biopsy for Diagnosis and Management of Biliary Tract Cancers
Brief Title: A Cell-free DNA Methylation Blood-Based Test for Biliary Tract Cancers Screening
Status: Recruiting | Type: Observational
Sponsor: Yingbin Liu, MD, PhD, FACS (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Xijing Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); West China Hospital (Other); Sun Yat-sen University (Other); Hunan Provincial People's Hospital (Other); Fudan University (Other)
Responsible Party: Sponsor-Investigator, Yingbin Liu, MD, PhD, FACS, principal investigator, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: BTC_ctDNAm_LYB_2025
Record Dates: First submitted 2025-09-10; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Gall Bladder Cancer; Intrahepatic Cholangiocarcinoma (Icc); Extrahepatic Cholangiocarcinoma; Hilar Cholangiocarcinoma; Billiary Track Cancer; ctDNA
Keywords: ctDNA methylation; Early diagnosis; Liquid biopsy; Billiary Track Cancer
MeSH Terms: conditions — Gallbladder Neoplasms; Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension; Klatskin Tumor; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- control（Internal training and validation sets）: Healthy individuals Patients with pathologically confirmed benign biliary lesions Patients with other gastrointestinal malignancies
- malignant（Internal training and validation sets）: patients with intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer
- malignant (Independent validation set): patients with suspected biliary tract malignancies
- control (Independent validation set): Healthy individuals

SUMMARY:
Biliary tract carcinoma (BTC), including gallbladder cancer, intrahepatic cholangiocarcinoma, and extrahepatic cholangiocarcinoma, ranks sixth in incidence among gastrointestinal malignancies and tenth in cancer-related mortality worldwide. Due to the lack of specific early symptoms, high malignancy, and frequent recurrence and metastasis, the rate of curative resection is only about 16.5%, and the overall 5-year survival rate is less than 5%. Early and accurate detection is therefore critical for improving patient outcomes. Circulating tumor DNA (ctDNA), a fraction of circulating free DNA (cfDNA), carries genetic and epigenetic information from tumor cells and can be detected even at the early stages of cancer development. Among various liquid biopsy biomarkers, ctDNA methylation shows particular advantages in sensitivity and specificity for early cancer detection and monitoring. This study aims to evaluate the application of cfDNA methylation liquid biopsy in the diagnosis and management of BTC.

DETAILED DESCRIPTION:
Biliary tract carcinoma (BTC), encompassing gallbladder cancer, intrahepatic cholangiocarcinoma, and extrahepatic cholangiocarcinoma, is an aggressive malignancy with poor prognosis. Globally, it ranks sixth in incidence among gastrointestinal cancers and tenth in cancer-related mortality. BTC is characterized by the absence of specific early symptoms, high degree of malignancy, and a strong tendency for recurrence and metastasis. The curative resection rate remains around 16.5%, and the overall 5-year survival rate is less than 5%.

Biliary tract inflammation (such as cholangitis, acute cholecystitis, sclerosing cholangitis, and autoimmune cholangitis) can lead to abnormal CA19-9 elevation. In addition, IgG4-related sclerosing cholangitis often affects elderly patients and may mimic hilar cholangiocarcinoma, creating diagnostic challenges. Imaging alone often lacks accuracy in differentiating benign from malignant biliary lesions, resulting in misdiagnosis and inappropriate clinical decision-making. The number of patients with incidentally detected BTC during surgery is rapidly increasing, and reoperations impose substantial trauma and socioeconomic burden.

Circulating tumor DNA (ctDNA) refers to DNA fragments released into the bloodstream from tumor cells through apoptosis, necrosis, or secretion. ctDNA carries genomic alterations (point mutations, indels, CNVs, fusions), epigenetic modifications (DNA methylation [5mC], hydroxymethylation [5hmC]), and structural features (fragment length, fragmentation patterns). Circulating free DNA (cfDNA) represents the total extracellular DNA in plasma or serum, of which ctDNA accounts for less than 1%. Accumulating evidence shows that ctDNA is detectable in the early stages of tumorigenesis, highlighting its clinical potential in early detection, diagnosis, treatment guidance, and post-treatment monitoring.

The choice of biomarker type is key to liquid biopsy applications, and ctDNA methylation offers distinct advantages. Liquid biopsy analytes include circulating tumor cells (CTCs), ctDNA, exosomes, and microRNAs (miRNAs), each with unique detection characteristics. ctDNA, directly derived from tumor cells, provides relatively high sensitivity for early detection and is currently the most widely used target in clinical practice. Research on ctDNA has focused mainly on methylation, somatic mutations, and copy number variations. Among these, ctDNA methylation balances both signal abundance and signal strength, offering clear advantages over other approaches. Methylation analysis methods include restriction enzyme digestion, affinity enrichment, and bisulfite conversion. Among them, bisulfite-based approaches are the most established and widely used.

Therefore, the application of cfDNA methylation liquid biopsy in BTC for early screening, differential diagnosis, prognostic monitoring, and therapeutic guidance holds great significance for improving diagnosis, treatment, and patient outcomes.

ELIGIBILITY:
Inclusion Criteria Internal Training and Validation Cohorts

* BTC patients

  1. Willing to voluntarily participate and able to comply with study procedures; if unable to read or sign, informed consent must be signed by a legally authorized representative (LAR).
  2. Age 18-80 years (inclusive).
  3. Able to provide required blood samples.
  4. Pathologically confirmed biliary tract carcinoma (TNM stage I-IV).
  5. Stable vital signs; ECOG performance status 0-1.
  6. Adequate organ function: AST/ALT ≤ 5 × ULN; Child-Pugh class A or B; WBC > 3 × 10⁹/L; ANC ≥ 1.5 × 10⁹/L; Platelets ≥ 75 × 10⁹/L; Hemoglobin ≥ 90 g/L; Creatinine clearance ≥ 60 mL/min; Total bilirubin ≤ 3 × ULN.
* Other gastrointestinal malignancies (to exclude BTC non-specific signals)

  1. Voluntary participation with signed informed consent (or by LAR).
  2. Age 18-80 years (inclusive).
  3. Able to provide required blood samples.
  4. Pathologically confirmed gastrointestinal malignancies other than BTC, including hepatocellular carcinoma, gastric cancer, colorectal cancer, and pancreatic cancer (TNM stage I-IV).
  5. Stable vital signs; ECOG performance status 0-1.
* Non-cancer participants (benign biliary disease)

  1. Able to provide written informed consent.
  2. Able to provide required blood samples.
  3. Age 18-80 years (inclusive).
  4. Pathologically or clinically diagnosed benign biliary diseases, including cholecystitis, cholelithiasis, choledocholithiasis, adenomyomatosis, gallbladder polyps, xanthogranulomatous cholecystitis, or primary sclerosing cholangitis.

External Validation Cohorts

* BTC patients

  1. Voluntary participation with signed informed consent (or by LAR).
  2. Imaging findings of malignant biliary stricture or mass, or serum CA19-9 > 100 U/mL, highly suspicious for BTC, with planned surgery or biopsy for pathological confirmation.
  3. Age 18-80 years (inclusive).
  4. Able to provide required blood samples.
  5. Stable vital signs; ECOG performance status 0-1.
  6. Adequate organ function: AST/ALT ≤ 5 × ULN; Child-Pugh class A or B; WBC > 3 × 10⁹/L; ANC ≥ 1.5 × 10⁹/L; Platelets ≥ 75 × 10⁹/L; Hemoglobin ≥ 90 g/L; Creatinine clearance ≥ 60 mL/min; Total bilirubin ≤ 3 × ULN.
* Healthy volunteers

  1. Able to provide written informed consent.
  2. Able to provide required blood samples.
  3. Age 18-80 years (inclusive).

Exclusion Criteria Training and Validation Cohorts

* Cancer patients

  1. Pregnant or breastfeeding women.
  2. History of organ transplantation or prior allogeneic bone marrow/stem cell transplantation.
  3. Blood transfusion within 7 days prior to blood collection.
  4. History of curative cancer treatment within 3 years prior to blood collection.
  5. Use of anti-tumor drugs within 30 days prior to blood collection.
  6. Known bleeding disorders.
  7. Known autoimmune diseases.
  8. Concurrent other malignancies or multiple primary tumors.
* Non-cancer participants

  1. Pregnant or breastfeeding women.
  2. History of organ transplantation or prior allogeneic bone marrow/stem cell transplantation.
  3. Blood transfusion within 7 days prior to blood collection.
  4. History of any malignant tumor.
  5. Known bleeding disorders.
  6. Known autoimmune diseases.
  7. Clinically significant abnormalities on routine examination (excluding hepatitis, hepatic cysts, or benign pulmonary nodules).

External Validation Cohorts

* Cancer patients

  1. Pregnant or breastfeeding women.
  2. History of organ transplantation or prior allogeneic bone marrow/stem cell transplantation.
  3. Blood transfusion within 7 days prior to blood collection.
  4. History of or ongoing curative cancer treatment within 3 years prior to blood collection.
  5. Use of anti-tumor drugs within 30 days prior to blood collection.
  6. Known bleeding disorders or autoimmune diseases.
  7. Concurrent other malignancies (including multiple primaries) or known cancer susceptibility gene carriers.
  8. Pathology confirmed benign disease after biopsy/surgery.
  9. Failure to confirm malignancy by pathology or imaging within 42 days after blood collection, or unclear lesion site/evidence.
  10. Special exclusion criteria:
* Pathology confirmed precancerous lesions.
* Any local/regional or systemic anti-tumor therapy (including surgery, radiotherapy, targeted therapy, or immunotherapy) prior to blood collection.
* Healthy volunteers

  1. Pregnant or breastfeeding women.
  2. History of organ transplantation or prior allogeneic bone marrow/stem cell transplantation.
  3. Blood transfusion within 7 days prior to blood collection.
  4. History of any malignant tumor.
  5. Known bleeding disorders or autoimmune diseases.
  6. Clinically significant abnormalities on health examination (excluding hepatitis, hepatic cysts, or benign pulmonary nodules).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprises individuals meeting inclusion criteria and not meeting any exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-03-21 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of the ctDNA methylation model in biliary tract cancer | Baseline
  Evaluate the overall sensitivity, specificity, and accuracy of the ctDNA methylation liquid biopsy model in the diagnosis of biliary tract cancer (BTC).

SECONDARY OUTCOMES:
Subtype-specific diagnostic performance | Baseline
  Sensitivity, specificity, and accuracy of the ctDNA methylation model in gallbladder cancer, intrahepatic cholangiocarcinoma, and extrahepatic cholangiocarcinoma.
Stage-specific diagnostic performance | Baseline
  Sensitivity, specificity, and accuracy of the model across BTC stages I-IV (TNM staging).
Differential diagnosis | Baseline
  Sensitivity, specificity, and accuracy of the ctDNA methylation model in distinguishing BTC from benign biliary lesions.

OTHER OUTCOMES:
Progression-Free Survival (PFS) | From date of diagnosis until documented progression or death, whichever occurs first, up to 5 years.
  To assess the association between ctDNA methylation and PFS in BTC patients.
Overall Survival (OS) | From date of diagnosis until death from any cause, up to 5 years.
  To assess the association between ctDNA methylation and OS in BTC patients.
Recurrence monitoring performance | Up to 5 years post-treatment
  Sensitivity and specificity of ctDNA methylation for monitoring recurrence and progression of biliary tract malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Yingbin Liu, PhD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chung DC, Gray DM 2nd, Singh H, Issaka RB, Raymond VM, Eagle C, Hu S, Chudova DI, Talasaz A, Greenson JK, Sinicrope FA, Gupta S, Grady WM. A Cell-free DNA Blood-Based Test for Colorectal Cancer Screening. N Engl J Med. 2024 Mar 14;390(11):973-983. doi: 10.1056/NEJMoa2304714. PMID 38477985
- [Background] Nagino M, Hirano S, Yoshitomi H, Aoki T, Uesaka K, Unno M, Ebata T, Konishi M, Sano K, Shimada K, Shimizu H, Higuchi R, Wakai T, Isayama H, Okusaka T, Tsuyuguchi T, Hirooka Y, Furuse J, Maguchi H, Suzuki K, Yamazaki H, Kijima H, Yanagisawa A, Yoshida M, Yokoyama Y, Mizuno T, Endo I. Clinical practice guidelines for the management of biliary tract cancers 2019: The 3rd English edition. J Hepatobiliary Pancreat Sci. 2021 Jan;28(1):26-54. doi: 10.1002/jhbp.870. Epub 2020 Dec 23. PMID 33259690
- [Background] Yang M, Zhao Y, Li C, Weng X, Li Z, Guo W, Jia W, Feng F, Hu J, Sun H, Wang B, Li H, Li M, Wang T, Zhang W, Jiang X, Zhang Z, Liu F, Hu H, Wu X, Gu J, Yang G, Li G, Zhang H, Zhang T, Zang H, Zhou Y, He M, Yang L, Wang H, Chen T, Zhang J, Chen W, Wu W, Li M, Gong W, Lin X, Liu F, Liu Y, Liu Y. Multimodal integration of liquid biopsy and radiology for the noninvasive diagnosis of gallbladder cancer and benign disorders. Cancer Cell. 2025 Mar 10;43(3):398-412.e4. doi: 10.1016/j.ccell.2025.02.011. PMID 40068597
- [Background] Vogel A, Bridgewater J, Edeline J, Kelley RK, Klumpen HJ, Malka D, Primrose JN, Rimassa L, Stenzinger A, Valle JW, Ducreux M; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Biliary tract cancer: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2023 Feb;34(2):127-140. doi: 10.1016/j.annonc.2022.10.506. Epub 2022 Nov 10. No abstract available. PMID 36372281